CLINICAL TRIAL: NCT00536952
Title: A Pilot Study of Pulmozyme (rhDNase) in Patients With Head and Neck Cancers Treated With Radiation and Chemotherapy
Brief Title: Pilot Study of Pulmozyme (rhDNase) in Patients With Head and Neck Cancers Treated With Radiation Therapy + Chemotherapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NU 06N2; STU00001045 (Other: Northwestern University IRB); GENENTECH-NU-06N2 (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — dornase alfa; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Pulmozyme
  Interventions: Drug: Pulmozyme; Radiation: Radiation Therapy
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Pulmozyme — Pulmozyme 2.5 mL ampules (2.5 mg) will be nebulized and inhaled once daily using a recommended nebulizer
  Other Names: dornase alfa inhalation solution
  Arms: Arm 1
Drug: Placebo — Placebo 2.5 mL ampules (2.5 mg) will be nebulized and inhaled once daily using a recommended nebulizer
  Arms: Arm 2
Radiation: Radiation Therapy — 5 days per week for 4 weeks

SUMMARY:
RATIONALE: Nebulized dornase alfa inhalation solution may decrease the thickness of saliva in the mouth and improve quality of life in patients undergoing radiation therapy and chemotherapy for head and neck cancer. It is not yet known whether dornase alfa inhalation solution is more effective than a placebo in lessening the discomfort of treatment in these patients.

PURPOSE: This randomized clinical trial is studying how well dornase alfa inhalation solution works compared with a placebo in treating patients with stage III or stage IV head and neck cancer undergoing radiation therapy and chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if use of nebulized dornase alfa inhalation solution can improve the overall daily symptom and quality of life as well as reduce treatment discomfort during radiotherapy and chemotherapy in patients with stage III or IV squamous cell carcinoma of the head and neck.
* To determine if once daily nebulized dornase alfa inhalation solution given prior to radiotherapy can reduce thick oropharyngeal secretions associated with curative radiotherapy and chemotherapy in these patients.
* To determine if reduction in thick oropharyngeal secretions with the use of nebulized dornase alfa inhalation solution can decrease the incidence of mucositis, infections, and aspiration pneumonia.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive nebulized dornase alfa inhalation solution via oral inhalation approximately 30 minutes prior to radiation therapy on days 1-5. Treatment continues for up to 4 weeks (weeks 3-6 of radiation therapy) in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive nebulized placebo via oral inhalation approximately 30 minutes prior to radiation therapy on days 1-5. Treatment continues for up to 4 weeks as in arm I.

All patients are assessed for treatment-related symptoms and treatment disturbance daily during radiation therapy. Patients are assessed for quality of life weekly during radiation therapy and then monthly during follow-up for 3 months. Clinical symptoms (i.e., mucositis, bacterial and fungal infections, and aspiration pneumonia) are also assessed weekly during radiation therapy.

Sputum samples are collected prior to initiating radiation therapy (at baseline) and periodically during week 3 of radiation treatment and evaluated for salivary DNA levels.

After completion of study therapy, patients are followed monthly for 3 months and then every 3-4 months for a minimum of 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, nasopharynx, oropharynx, hypopharynx, or larynx

  * Stage III or IV disease
  * Confirmation from primary site and/or lymph nodes
* Patients with a history of head and neck cancer allowed provided they have not received prior radiotherapy

  * Prior localized radiotherapy for skin cancer arising in the head and neck region is allowed
* Planning to receive radiation therapy and chemotherapy to the head and neck regions with a minimum expected radiation dose of 60 Gy over 6 weeks

  * Chemotherapy may include but is not limited to, cisplatin or carboplatin, fluorouracil, hydroxyurea, docetaxel, and/or cetuximab

    * Induction chemotherapy allowed

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* No prior allergic reaction or known sensitivity to dornase alfa inhalation solution
* No significant active infection or other severe complicating medical illness
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent amifostine
* No mouth wash 1 hour before or after dornase alfa inhalation solution administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-02; Primary Completion 2014-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-related symptoms as assessed daily by the Head and Neck Symptom Inventory Scale (MD Anderson Symptom Inventory) | 5 times per week during study treatment and once per month up to 3 months post-treatment
Quality of life as assessed weekly by the Functional Assessment of Cancer Therapy - Head & Neck Neck questionnaire | Weekly during study treatment and once per month up to 3 months post-treatment.
Patient comfort and/or disturbance during radiotherapy treatment as assessed daily by Radiation Treatment Disturbance Disturbance Measures questionnaire | Daily during radiation treatment

SECONDARY OUTCOMES:
Reduction in amount of thick oropharyngeal secretions associated with cancer therapy. | At baseline, prior to radiation and study treatment, and after radiation.
Incidence of mucositis, infections, and aspiration pneumonia | Weekly during study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bharat B. Mittal, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States